CLINICAL TRIAL: NCT01841151
Title: Does Neurofeedback and Working Memory Training Improve Core Symptoms of ADHD in Children and Adolescents? A Comparative, Randomized and Controlled Study.
Brief Title: Neurofeedback and Working Memory Training for Children and Adolescents With ADHD
Acronym: KITE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Region Stockholm (Other Government); Child and Adolescent Psychiatry, Stockholm (Industry); Stiftelsen Sunnerdahls Handikappfond (Other); Swedish Foundation for Strategic Research (Other)
Responsible Party: Principal Investigator, Sven Bölte, Professor, PhD, head of pediatric neuropsychiatry unit, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KITE
Record Dates: First submitted 2013-04-20; First posted 2013-04-26 (Estimated); Results first posted 2025-08-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Attention Deficit Disorder
Keywords: AD/HD in Children and Adolescents
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- SCP training (Active Comparator): Neurofeedback 1 (NF1) Slow Cortical Potential (SCP) training
  Interventions: Behavioral: SCP training
- Live Z-score training (Active Comparator): Neurofeedback 2 (NF2) Live Z-score training
  Interventions: Behavioral: Live Z-score training
- WM training (Active Comparator): Working Memory training (WMt)
  Interventions: Behavioral: WM training
- Waiting-list (No Intervention): Treatment as usual only

INTERVENTIONS:
Behavioral: SCP training
  Arms: SCP training
Behavioral: Live Z-score training
  Arms: Live Z-score training
Behavioral: WM training
  Arms: WM training

SUMMARY:
The purpose of this study is to investigate if neurofeedback and working memory training improves core symptoms of ADHD in children and adolescents.

DETAILED DESCRIPTION:
This study investigates two types of Neurofeedback (NF), one well-established and well-researched protocol called Slow Cortical Potential NF (SCP), and a newer and less researched, yet popular among private clinicians, the so-called live z-score training (LZT). These methods are compared to working memory training (WMT) and a passive control condition, treatment-as-usual only (TAU). The active conditions (SCP/LZT/WMT) are delivered high frequent, with 5 sessions/week, for a total of 25 sessions.

Outcomes measures are taken at Preintervention and Postintervention, as well as at a 6-month follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

* Clinical AD/HD diagnose according to DSM-IV-TR and K-SADS interview, 9-17 years old, unmedicated or under stable medication with stimulants or corresponding since at least one month.

Exclusion Criteria:

* IQ <70 (WISC-IV or WAIS-IV), clinically instable psychiatric state e.g. severe depression, OCD, self-injurious behaviour, bipolar disorder, severe somatic (neurologic) disease, very limited knowledge in the Swedish language.

Ages: 9 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 202 (Actual)
Dates: Start 2013-08 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2020-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sven Bölte, Professor, Principal Investigator — Karolinska Institute, Competence Center of Neurodevelopmental Disorders (KIND)
Locations (1):
- Cap Bup-Kind, Stockholm, Sweden

REFERENCES:
- [Background] Hasslinger, J., Sirviö, S., Berggren, S., Myers, L., Flygare, O., Tammimies, K., & Bölte, S. (2016). A comparative randomized controlled pragmatic trial of neurofeedback and working memory training for children with attention-deficit/hyperactivity disorder: protocol. Translational Developmental Psychiatry, 4(1). https://doi.org/10.3402/tdp.v4.30556
- [Result] Hasslinger J, D'Agostini Souto M, Folkesson Hellstadius L, Bolte S. Neurofeedback in ADHD: A qualitative study of strategy use in slow cortical potential training. PLoS One. 2020 Jun 4;15(6):e0233343. doi: 10.1371/journal.pone.0233343. eCollection 2020. PMID 32497051
- [Result] Hasslinger J, Bolte S, Jonsson U. Slow Cortical Potential Versus Live Z-score Neurofeedback in Children and Adolescents with ADHD: A Multi-arm Pragmatic Randomized Controlled Trial with Active and Passive Comparators. Res Child Adolesc Psychopathol. 2022 Apr;50(4):447-462. doi: 10.1007/s10802-021-00858-1. Epub 2021 Sep 3. PMID 34478006
- [Result] Hasslinger J, Jonsson U, Bolte S. Immediate and Sustained Effects of Neurofeedback and Working Memory Training on Cognitive Functions in Children and Adolescents with ADHD: A Multi-Arm Pragmatic Randomized Controlled Trial. J Atten Disord. 2022 Sep;26(11):1492-1506. doi: 10.1177/10870547211063645. Epub 2022 Jan 16. PMID 35034510
- See also: Competence Center of Neurodevelopmental Disorders (KIND) — https://ki.se/kind/center-of-neurodevelopmental-disorders-at-karolinska-institutet-kind
- See also: Webpage for BUP KIND - the KITE-project — http://ki.se/en/kind/kite-neurofeedback-and-working-memory-training

RESULTS

PARTICIPANT FLOW:
Groups:
- SCP Training: Neurofeedback 1 (NF1) Slow Cortical Potential (SCP) training
  SCP training
- Live Z-score Training: Neurofeedback 2 (NF2) Live Z-score training (LZT)
  Live Z-score training
- WM Training: Working Memory training (WMt)
  WM training
Period: Overall Study
Arm/Group | SCP Training | Live Z-score Training | WM Training | Waiting-list
Started | 51 | 50 | 51 | 50
Completed | 43 | 46 | 42 | 49
Not Completed | 8 | 4 | 9 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SCP Training | Live Z-score Training | WM Training | Waiting-list | Total
Number analyzed (Participants) | 51 | 50 | 51 | 50 | 202
Age, Continuous [Mean (Full Range); unit: years]
  Range | 12.35 [9 to 18] | 12.41 [9 to 17] | 12.61 [9 to 18] | 12.21 [9 to 17] | 12.40 [9 to 18]
Age, Customized [Mean (Standard Deviation); unit: years]
  Mean (Sd) | 12.35 (2.65) | 12.41 (2.30) | 12.61 (2.74) | 12.21 (2.41) | 12.40 (2.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 13 | 9 | 14 | 49
  Male | 38 | 37 | 42 | 36 | 153
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Symptom Severity - Conners3 ADHD-index [Mean (Standard Deviation); unit: units on a scale] — Conners-3, ADHD-index, T-scores Scores range from 40-90 (swedish norms) Higher score indicate greater symptom severity.
  units on a scale
    Conners-3 Self-rating | 69.24 (16.15) | 67.12 (15.15) | 72.26 (16.67) | 70.06 (15.79) | 69.67 (15.94)
    Conners-3 Parent-rating | 80.51 (13.91) | 82.84 (9.16) | 81.32 (12.85) | 82.84 (10.91) | 81.86 (11.82)
    Conners-3 Teacher-rating | 62.76 (13.37) | 65.83 (14.88) | 64.27 (15.47) | 66.67 (14.61) | 64.92 (14.55)
Symptom Severity (Range) [Median (Full Range); unit: units on a scale] — Conners-3, adhd-index, T-scores Scores range from 40-90 (swedish norms)
  units on a scale
    Self-Rating | 67 [46 to 90] | 62.5 [46 to 90] | 72.5 [45 to 90] | 72 [46 to 90] | 69 [45 to 90]
    Parent-Rating | 89 [46 to 90] | 88.5 [61 to 90] | 89 [46 to 90] | 89 [47 to 90] | 89 [46 to 90]
    Teacher-Rating | 59 [44 to 90] | 65 [43 to 90] | 65 [43 to 90] | 67 [44 to 90] | 64 [43 to 90]

OUTCOME MEASURES:

1. Primary Outcome: Conners 3 ADHD-index
Description: Presented below are the within-group differences from baseline to 6-month follow up, for the ADHD-index of the Conners-3.
  Positive numbers indicate symptom improvements.
  *The ADHD-index raw score can range from 0-20, with higher score indicating greater symptom severity. The Reliable Change Index (RCI) is 2.88.
Time Frame: Up to seven months
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | SCP Training | Live Z-score Training | WM Training | Waiting-list
Number analyzed (Participants) | 51 | 50 | 51 | 50
score on a scale
  Conners3-ADHD-index Self-rating | 1.21 [0.12 to 2.29] | 1.37 [0.26 to 2.47] | 1.44 [0.53 to 2.36] | 0.78 [-0.13 to 1.70]
  Conners3-ADHD-index Parent-rating | 1.81 [0.48 to 3.14] | 2.26 [0.75 to 3.78] | 2.22 [1.07 to 3.37] | 0.60 [-0.47 to 1.67]
  Conners3-ADHD-index Teacher-rating | 1.32 [-0.28 to 2.93] | 3.37 [1.78 to 4.95] | 2.80 [1.06 to 4.54] | -0.66 [-2.12 to 0.79]

ADVERSE EVENTS:
Time Frame: Adverse Events were monitored using the Pediatric Side Effects Checklist (Pavuluri & Janicak, 2004) during the five-week training period. Additionally adverse events were assessed during the baseline-assessment (week 0), at the post-assessment (week 7) and at the follow-up assessment (6-month after post-assessment).
Groups:
- Live Z-score Training: Neurofeedback 2 (NF2) Live Z-score training
  Live Z-score training
Arm/Group | SCP Training | Live Z-score Training | WM Training | Waiting-list
All-Cause Mortality (participants affected / at risk) | 0/51 | 0/50 | 0/51 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/51 | 0/50 | 0/51 | 0/50
Other Adverse Events (participants affected / at risk) | 0/51 | 0/50 | 0/51 | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-06-07): https://cdn.clinicaltrials.gov/large-docs/51/NCT01841151/Prot_SAP_000.pdf